CLINICAL TRIAL: NCT06135987
Title: Clinical Evaluation of URGOSTART PLUS® BORDER, URGOSTART PLUS® PAD and URGOSTART INTERFACE® in the Local Treatment of Diabetic Foot Ulcers and Venous Leg Ulcer of Mixed Etiology : French Prospective and Multicentric Observational Study
Brief Title: Clinical Evaluation in Real Life of TLC-NOSF Dressings in the Local Treatment of Chronic Wounds (DFU and VLU)
Acronym: STARTLIFE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A02414-37
Record Dates: First submitted 2023-10-16; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Real Life Study; TLC-NOSF Dressings; Venous Leg Ulcer; Diabetic Foot Ulcer; QoL Questionnaire
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TLC-NOSF dressings (D'URGOSTART PLUS® BORDER, URGOSTART PLUS® PAD and URGOSTART INTERFACE®) — Clinical evaluation of the dressing in the local treatment of chronic wounds (DFU and VLU)

SUMMARY:
The objective of this study is to document the performance and the safety of UrgoStart Plus® Border, UrgoStart Plus® Pad and UrgoStart Interface® in the local treatment of diabetic foot ulcers (neuropathic or neuroischemic - non-critical ischemia) and venous or mixed predominantly venous leg ulcers, in real life conditions and current practice, in France.

DETAILED DESCRIPTION:
This is an observational, non-interventional, prospective multicenter study, carried out in real-life conditions on CE marked medical devices used for their intended purpose.

The study will be carried out in France, in accordance with national and European regulations (RDM 2017/745).

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatient having signed informed consent
* Patient with a venous leg ulcer (VLU) Or with a diabetic foot ulcer (DFU)
* Prescription of one of the 3 dressings: UrgoStart Plus® Border, UrgoStart Plus® pad or UrgoStart Interface®
* Patient can be followed over 12 weeks by the investigator, according to his/her practices
* Patient able to participate in the study and complete a self-questionnaire without difficulty

Exclusion Criteria:

* Hemorrhagic wound
* Cancerous wound
* Fistulous wound revealing a deep abscess
* Presence of dry necrosis partially or completely covering the wound bed
* Infected wound
* Osteitis
* Critical or acute ischemia
* Patient for whom a surgical procedure related to the treated wound is scheduled within 12 weeks following the inclusion visit
* Patient with known sensitivity to one of the studied dressings components
* Pregnant or breastfeeding patient
* Patient under the protection of justice or under guardianship or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients participating in this clinical evaluation suffering of:
  * a predominantly venous or mixed leg ulcer,
  * or a neuropathic or neuroischemic diabetic foot ulcer (without critical ischemia) that the investigating physician has decided to treat with one or other of the 3 following dressing containing TLC-NOSF : UrgoStart Plus® Border, UrgoStart Plus® Pad or UrgoStart Interface®
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complete healed chronic wound (venous leg ulcer and Diabetic foot ulcer) at 12 weeks | 12 weeks
  Complete ulcer closure (100% re-epithelialization) over 12 weeks of treatment with UrgoStart Plus® Border, UrgoStart Plus® pad and UrgoStart Interface® dressings

SECONDARY OUTCOMES:
Time to wound closure | 12 weeks
  For healed patients: time to wound closure (in days)
Relative reduction in wound surface area | 12 weeks
  Relative reduction in wound surface area (in %) during intermediate and final visits
EQ5D5L quality of life questionnaire | 12 weeks
  The evolution of the patient quality of life assessed with the EuroQoL 5D-5L will be evaluated between baseline and at last visit.
Tolerance : the nature and number of adverse event related to the use of the testing dressings | 12 weeks
  The nature and number of adverse event related to the use of the testing dressings (UrgoStart Plus® Border, UrgoStart Plus® pad and UrgoStart Interface® dressings) (serious/ non-serious) will be described.
Defectuosity of the device | 12 weeks
  Description of the defects of the devices used.

CONTACTS AND LOCATIONS:
Locations (1):
- Pr Agnès HARTEMANN, Paris, France